CLINICAL TRIAL: NCT05246774
Title: Study of Serum and Urinary Biomarkers and Radiation Cystitis in Patients Treated With Radiotherapy for Localized Prostate Cancer
Acronym: RABBIO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2021PPRC09; 2021-A03196-35 (Other: IDRCB)
Record Dates: First submitted 2022-02-09; First posted 2022-02-18 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Radiation Cystitis; Prostate Cancer; Radiotherapy Side Effect
MeSH Terms: conditions — Prostatic Neoplasms; Radiation Injuries | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Several samples will be collected :
  * fecal samples
  * urine samples
  * blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Biological sample collection — The following biological samples will be collected on 4 occasions (at enrollment, 4 weeks after, 12 weeks after and 52 weeks after) :
  * fecal sample
  * urinary sample
  * blood sample (22 ml at each occasion)
Other: Questionnaires — The following questionnaires will be filled by the patients on 4 occasions (at enrollment, 4 weeks after, 12 weeks after and 52 weeks after) :
  * CTCAE Radiation Adverse Event Questionnaire
  * Lower Urinary Tract Disorders Questionnaire (IPSS Score)
  * Quality of Life Questionnaire (FACT-P)
  * Physical Activity Questionnaire (IPAQ)

SUMMARY:
Prostate cancer represents the 1st diagnosed cancer in men, with 50400 new cases and 8100 deaths in 2018. Improved diagnostic and therapeutic strategies have led to a 3.7% decrease in mortality between 2010 and 2018 with a 5- and 10-year survival rate of 93% and 80%, respectively.

Pelvic conformal radiotherapy is an important therapeutic technique in the management of pelvic cancers, particularly prostate cancer. However, despite the improvement in radiation techniques, this technique is responsible for acute and late adverse events at the bladder level, these symptoms being grouped under the term radiation cystitis. It has a clear impact on the quality of life of patients. Acute radiation cystitis is likely to occur during treatment or within 3 months after radiotherapy. Its incidence is estimated at nearly 50%. The late form appears on average 2 years after radiation, but can sometimes occur 10 or 20 years later. Its incidence is 5 to 10% of cases.

Although certain factors have been identified, such as the dose received, fractionation or comorbidities, the pathophysiology of radiation-induced cystitis remains unclear, particularly because of the risks of complications arising from access to bladder tissue post-irradiation, thus limiting our knowledge as well as the therapies targeting this process. The use of biomarkers in liquid biopsies allows us to understand the problem of access to irradiated tissues and to highlight protein changes, prognostic of radiation-induced visceral toxicity.

Few works are published on the evaluation of inflammatory and pro-fibrotic biomarkers of radiation-induced cystitis in liquid biopsies. Only 2 retrospective studies have shown a correlation between late radiation cystitis and increased levels of plasminogen activator inhibitor 1 (PAI-1), matrix metalloproteinase inhibitors (TIMP1 and TIMP2), hepatocyte growth factor (HGF), vascular endothelial growth factor (VEGF) and placental growth factor (PIGF) in urine. However, none of these studies explored the variation of biomarkers in the early stage of radiation-induced bladder toxicity.

This would suggest the feasibility of prospective assay of overexpression of these proteins in liquid biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate;
* Localized adenocarcinoma of the prostate according to the D'Amico Risk Classification for Prostate Cancer;
* Eligible for external beam radiation therapy and/or brachytherapy;
* Patient able, in the opinion of the physician-investigator, to communicate well, understand and comply with the requirements of the study;
* Patient with a phone or a computer.

Exclusion Criteria:

* Patient with advanced or metastatic prostate cancer;
* Patient receiving pre-irradiation hormone therapy;
* Patient with bladder or urethral cancer or a history of it;
* Previous urinary tract surgery (bladder augmentation, cystectomy);
* Patient participating in an interventional clinical study;
* Patient with a history of pelvic irradiation;

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is composed of adult men with localized prostate cancer who are eligible for radiation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Concentration of 33 urinary and serum biomarkers potentially related to radiation cystitis between enrollment and 12 weeks after the start of radiotherapy. | Up to to 12 weeks after the start of radiotherapy
  The change in expression of the 33 inflammatory and remodeling biomarkers will be assessed by :
  * the MILLIPLEX® MAP technique for the analysis of circulating markers
  * the flow cytometry method for the analysis of the immune population.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital d'Instruction des Armées Bégin, Saint-Mandé, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Helissey C, Cavallero S, Mondot S, Parnot C, Yssaad H, Becherirat S, Guitard N, Thery H, Schernberg A, Breitwiller H, Chargari C, Francois S. Correlation Between Serum and Urine Biomarkers and the Intensity of Acute Radiation Cystitis in Patients Treated With Radiation Therapy for Localized Prostate Cancer: Protocol for the Radiotoxicity Bladder Biomarkers (RABBIO) Study. JMIR Res Protoc. 2023 Jan 10;12:e38362. doi: 10.2196/38362. PMID 36626198